CLINICAL TRIAL: NCT02576379
Title: The Impact of a Helicopter Emergency Medical System on Prognosis in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kamilia S. Funder, MD., Rigshospitalet, Denmark
Other Study IDs: ALH3-KF-2015
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Thrombolysis
Keywords: Helicopter Emergency Medical System; Mortality; Labour market affiliation; Modified Rankin Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HEMS patients: Patients suspected of suffering from a vascular condition within the geographical area covered by both HEMS and GEMS, and were transported by Helicopter Emergency Medical System (HEMS) to the regional stroke unit at Copenhagen University Hospital Roskilde in a 36-month period from May 1st 2010 until April 30th 2013.
- GEMS patients: Patients suspected of suffering from a vascular condition within the geographical area covered by both HEMS and GEMS, and were transported by Ground Emergency Medical System (GEMS) to the regional stroke unit at Copenhagen University Hospital Roskilde in a 40-month period from January 1st 2010 until April 30th 2013.

SUMMARY:
Stroke is a leading cause of death and disability, and 15 million people suffer a stroke each year; one-third die and one-third are left permanently disabled. Because the risk of stroke increases with age, it has been considered a disease of the elderly, but stroke also occurs in middle-aged people.

Thrombolysis with tissue plasminogen activator (tPA) is the preferred choice of reperfusion therapy of ischemic stroke if performed within 4.5 hours from symptom onset. Time to thrombolysis is associated with improved outcome: the sooner the treatment, the less risk of serious - and possibly permanent - damage to the brain. Unfortunately, only a small fraction of stroke patients make it to thrombolysis within the 4.5-hour; one explanation may be system delays including prolonged transportation.

In May 2010, the first physician-staffed Helicopter Emergency Medical Service (HEMS) was implemented in the Eastern part of Denmark. An observational study evaluating the short-term effects of HEMS implementation compared patients transported by conventional ground ambulance (Ground Emergency Medical Service (GEMS)) to patients transported by HEMS. Patients transported by helicopter had increased time to specialized care. However, both 30-day and 1-year mortality was slightly lower in patients transported by HEMS, although not significant, as was the degree of disability at three months measured by the modified Rankin Scale (mRS).

ELIGIBILITY:
Inclusion Criteria:

* All patients arriving at the regional stroke unit at Copenhagen University Hospital, Roskilde, suspected of an acute vascular condition within the geographical area covered by both HEMS and GEMS in a 40-month period from January 1st 2010 until April 30th 2013.

Exclusion Criteria:

* For patients with multiple contacts; only the first contact is included in the data for analysis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients arriving at the regional stroke unit at Copenhagen University Hospital, Roskilde, suspected of an acute vascular condition within the geographical area covered by both HEMS and GEMS in a 40-month period from January 1st 2010 until April 30th 2013.
  The geographical catchment area is defined as the area from where HEMS transported patients the first year of implementation.
  We compare stroke patients transported by HEMS with stroke patients transported by GEMS.
Sampling Method: Probability Sample
Enrollment: 1068 (Actual)
Dates: Start 2010-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Risk of death during follow-up | 2 - 5.5 years after admission to the stroke unit.
  Mortality during the follow-up period will be analysed for differences between GEMS and HEMS. Follow-up period is until May 1st 2015. Because of varying access to information on covariates depending on the diagnosis and treatment of the patient, we conduct the analysis as follows: 1) the whole study population; adjusted for sex and age, 2) patients who were suspected of suffering from a vascular condition; adjusted for sex, age and comorbidity (defined as one of the following conditions; diabetes, atrial fibrillation, hypertension, previous myocardial infarction, and previous stroke), and 3) patients who underwent thrombolysis; adjustment for sex, age, comorbidity, and initial National Institutes of Health Stroke Scale (NIHSS) score.

SECONDARY OUTCOMES:
The risk of death at 30 day. | 30 days after admission to the stroke unit.
  Patients are divided into the same three sub-groups and adjusted for the same potential confounders as described in the primary outcome analysis.
Modified Rankin Scale (mRS) after three months. | Three months
  Assessed in patients who underwent thrombolysis.
The risk of involuntary early retirement during the follow-up period. | 2 - 5.5 years after admission to the stroke unit.
  Assessed in all patients suspected of suffering from a vascular condition between 18 and 60 years of age to ensure a sample that was at risk of involuntary early retirement during the full follow-up period.
The risk of reduced workability two years after the vascular event | Two years after admission to the stroke unit
  Assessed in all patients suspected of suffering from a vascular condition between 18 and 60 years of age to ensure a sample that was at risk of involuntary early retirement during the full follow-up period.
The percentage of time on social transfer payments during the first two years. | Two years after admission to the stroke unit
  Assessed in all patients suspected of suffering from a vascular condition between 18 and 60 years of age to ensure a sample that was at risk of involuntary early retirement during the full follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Kamilia S. Funder, MD, Principal Investigator — Department of Anesthesia, Center of Head and Orthopedics, section 4231, Copenhagen University Hospital, Rigshospitalet; Jacob Steinmetz, MD, PhD, Study Director — Department of Anesthesia, Center of Head and Orthopedics, section 4231, Copenhagen University Hospital, Rigshospitalet

REFERENCES:
- [Background] Wahlgren N, Ahmed N, Davalos A, Hacke W, Millan M, Muir K, Roine RO, Toni D, Lees KR; SITS investigators. Thrombolysis with alteplase 3-4.5 h after acute ischaemic stroke (SITS-ISTR): an observational study. Lancet. 2008 Oct 11;372(9646):1303-9. doi: 10.1016/S0140-6736(08)61339-2. Epub 2008 Sep 12. PMID 18790527
- [Background] Hesselfeldt R, Gyllenborg J, Steinmetz J, Do HQ, Hejselbaek J, Rasmussen LS. Is air transport of stroke patients faster than ground transport? A prospective controlled observational study. Emerg Med J. 2014 Apr;31(4):268-72. doi: 10.1136/emermed-2012-202270. Epub 2013 Feb 6. PMID 23389831
- [Derived] Funder KS, Rasmussen LS, Lohse N, Hesselfeldt R, Siersma V, Gyllenborg J, Wulffeld S, Hendriksen OM, Lippert FK, Steinmetz J. The impact of a physician-staffed helicopter on outcome in patients admitted to a stroke unit: a prospective observational study. Scand J Trauma Resusc Emerg Med. 2017 Feb 23;25(1):18. doi: 10.1186/s13049-017-0363-3. PMID 28231814